CLINICAL TRIAL: NCT04031001
Title: Vascular No-React Graft Against Infection
Acronym: VASC-REGAIN
Status: Completed | Type: Observational
Sponsor: Catharina Ziekenhuis Eindhoven (Other)
Responsible Party: Principal Investigator, Marc van Sambeek, prof. dr. M.R.H.M. van Sambeek, Catharina Ziekenhuis Eindhoven
Other Study IDs: NL59973.100.16
Record Dates: First submitted 2018-10-05; First posted 2019-07-24 (Actual); Last update posted 2023-12-21 (Actual); Status verified 2023-12

CONDITIONS: Vascular Infections

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: No-React Non-valved Conduit — Operative replacement of infected graft or implantation in infected area.

SUMMARY:
This study seeks to demonstrate the effectiveness and safety of the Non-valved Conduit for CE marking on the basis of infection. The rationale for infection resistance with the conduit is that BioIntegral Surgical No-React® treated products have a well-documented history of infection resistance in hybrid vascular settings.

ELIGIBILITY:
Inclusion Criteria:

* Infected prosthetic graft and/or bifurcation
* High risk of infection at graft implantation
* Mycotic aneurysm
* No alternative available

Exclusion Criteria:

* Below-knee procedure
* AV access

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with (a high risk for) infection.
Sampling Method: Probability Sample
Enrollment: 43 (Actual)
Dates: Start 2017-12-22 (Actual); Primary Completion 2021-02-06 (Actual); Study Completion 2021-07-13 (Actual)

PRIMARY OUTCOMES:
Percentage of graft infection 3 months after implantation | 3 months after implantation
  Percentage of graft infection 3 months after implantation as assessed with different infection parameters: CRP value, leukocytes, Samson classification of infection, temperature, wound healing, wound infection, purulence

SECONDARY OUTCOMES:
Percentage of patency 12 months after implantation | 12 months after implantation
  Percentage of patency 12 months after implantation as assessed with duplex ultrasound or CT imaging. <50% stenosis are defined as patent

CONTACTS AND LOCATIONS:
Locations (1):
- Catharina Ziekenhuis, Eindhoven, Netherlands